CLINICAL TRIAL: NCT06679673
Title: An Explorative Study of SHR-1701 Combined with SHR2554 and BP102(bevacizumab) for Metastatic Colorectal Cancer.
Brief Title: SHR-1701 Combined with SHR2554 and BP102 for MCRC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Xu, Prof., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-IIT-SHR1701-SHR2554-BP102
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — SHR-1701

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SHR-1701+BP102±SHR2554 (Experimental): The first 6 subjects will be treated with SHR-1701+BP102, and the subsequent subjects will be treated with SHR-1701+BP102+SHR2554
  Interventions: Drug: SHR-1701; Drug: BP102; Drug: SHR2554

INTERVENTIONS:
Drug: SHR-1701 — SHR-1701
Drug: BP102 — BP102
Drug: SHR2554 — SHR2554

SUMMARY:
Response to oncologic treatment in mCRC is currently limited.

DETAILED DESCRIPTION:
This is a single-center, open-labeled study exploring the efficacy and safety of SHR-1701 combined with SHR2554 and BP102 in the treatment of metastatic colorectal cancer (mCRC) .

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years;
* Histological confirmed metastatic colorectal cancer;
* ECOG PS 0-1;
* At least one measurable lesion (according to RECIST1.1);
* Adequate hepatic, renal, coagulation, and hematologic functions;
* Agree to use contraception during the study and 3 months after the end of the study. Negative serum pregnancy test at screening for women of childbearing potential;
* Patients voluntarily enroll in the study.

Exclusion Criteria:

* The patient has had other malignant tumors within 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* Symptomatic brain or meningeal metastases (except for those whose BMS disease is stable for at least 4 weeks);
* Allergy to the study drug or any of its excipients;
* Prior treatment with immune checkpoint inhibitors;
* Received the following treatments before the first study treatment;

  1. Major surgery within 28 days before treatment (tissue biopsy for diagnostic purposes is permitted).
  2. Prior use of immunosuppressive medications, excluding nasal and inhaled corticosteroids or physiologic doses of systemic steroids (i.e., no more than 10 mg/d prednisone or equivalent pharmacologic doses of other corticosteroids) within 7 days before treatment;
  3. Received immunomodulatory drugs within 3 weeks before treatment;
  4. Received live attenuated vaccine within 28 days before treatment;
  5. Receipt of other antitumor systemic therapy within 28 days prior to treatment;
* Presence of any active autoimmune disease or history of autoimmune disease with expected relapse;
* A known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
* Human immunodeficiency virus (HIV) infection or known AIDS, untreated active hepatitis, HBV-DNA ≥ 2500 IU/ml and abnormal liver function; hepatitis C or co-infection with hepatitis B and hepatitis C;
* A history of interstitial lung disease or non-infectious pneumonia, etc.;
* Within 6 months before enrollment, the following conditions: myocardial infarction, severe/unstable angina, NYHA class 2 or greater cardiac insufficiency, and clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention; hypertension with poorly controlled by medications;
* A history of severe bleeding within 3 months (>30 ml at a time) or hemoptysis within 1 month (>5 ml at a time) or a thromboembolic event (including pulmonary embolism, cerebral infarction, etc.) within 12 months;
* Surgical treatment (except biopsy) within 6 weeks or unhealed surgical incision;
* Long-standing unhealed wounds or fractures that have not healed properly
* Imaging showing that the tumor has invaded a vital vascular perimeter or if, in the judgment of the investigator, the patient's tumor has a very high likelihood of invading a vital blood vessel and causing a fatal hemorrhage during therapy
* A history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, or active gastrointestinal bleeding within 6 months before the first study treatment
* Urine routine showed urine protein ≥2+, and 24-hour urine protein level >1.0g;
* Unable to take the drug orally, or has a condition judged by the investigator to affect the absorption of the drug;
* Pregnancy, lactation, and unwillingness of reproductively active subjects to use effective contraception;
* Other conditions deemed by the investigator to be ineligible for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | assessed up to 1 year
  the proportion of patients with complete response or partial response, using RECIST v 1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | assessed up to 1 year
  the proportion of patients with complete response, partial response or stable disease, using RECIST v 1.1.
Progression-Free Survival (PFS) | assessed up to 1 year
  time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
Overall survival (OS) | assessed up to 2 year
  time from enrollment to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery Fudan University Shanghai Caner Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No